CLINICAL TRIAL: NCT05469061
Title: The Safety and Efficacy of Tislelizumab in Combination With Chemotherapy for Conversion Therapy of Locally Nonresectable ESCC，A Single-arm Study
Brief Title: Tislelizumab in Combination With Chemotherapy for Conversion Therapy of Locally Nonresectable ESCC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-SR-372
Record Dates: First submitted 2022-06-08; First posted 2022-07-21 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Esophageal Squamous Cell Carcinoma; Locally Advanced Carcinoma
Keywords: Drug: Tislelizumab; Chemotherapy
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — tislelizumab; Fluorouracil; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tislelizumab plus Chemotherapy (Experimental): In the single experimental arm, patients with locally nonresectable disease were subjected to receive neoadjuvant tislelizumab (200mg) plus chemotherapy (FP regimen) for conversion therapy. If conversion therapy succeeds, patients would proceed to surgery and adjuvant therapy. Otherwise, if patients were still not resectable after the conversion therapy, they will be treated by tislelizumab plus chemotherapy with or without palliative radiotherapy .
  Interventions: Drug: Tislelizumab; Drug: 5-FU; Drug: cis Platinum

INTERVENTIONS:
Drug: Tislelizumab — The 1st to 3rd doses were administered concurrently with FP regimen chemotherapy, 200 mg Tislelizumab each, on D1, D22 and D43 by intravenous infusion. In patients with successful conversion, one dose of 200 mg was administered 21 days after surgery in concurrent with the 4th to 6th cycles of 5-Fu, then 6 cycles of 200 mg Tislelizumab as adjuvant therapy; in patients with failed conversion, chemotherapy combined with tislelizumab were administered, with or without radiation therapy.
Drug: 5-FU — A FP regimen with 5-Fu 850mg/m^2 d1-4 + cis-platinum 850mg/m^2 d1-4 was used, on D1, D22 and D43 infused intravenously. 3 cycles of 5-Fu 850mg/m^2 d1-4 adjuvant chemotherapy were started at 21 days after surgery in patients with a successful conversion. In patients with failed conversion, chemotherapy combined with tislelizumab were administered, with or without radiation therapy.
Drug: cis Platinum — A FP regimen with 5-Fu 850mg/m^2 d1-4 + cis-platinum 850mg/m^2 d1-4 was used, on D1, D22 and D43 infused intravenously. In patients with failed conversion, chemotherapy combined with tislelizumab were administered, with or without radiation therapy.

SUMMARY:
This is a single-arm，open-label study to evaluate the efficacy and safety of tislelizumab plus chemotherapy for conversion therapy of patients with locally nonresectable ESCC.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 75 years;
2. Understand the research procedure and content, and voluntarily sign written informed consent;
3. Patients with clinical stage IIA-IIIB esophageal cancer were assessed by endoscopic ultrasonography, CT/MRI and other imaging.
4. Esophageal surgery experts believe that patients with potentially resectable esophageal cancer
5. No blood transfusion was received 3 months before enrollment;
6. ECOG PS score: 0-1.

Exclusion Criteria:

* Patients meeting any of the following criteria are not eligible for inclusion:

  1. Women who are pregnant or breastfeeding;
  2. previous or concurrent malignancy;
  3. Participated in clinical trials of other drugs within four weeks;
  4. Have a history of immune deficiency, or other acquired or congenital immune deficiency diseases, or have a history of organ transplantation, or have a history of serious chronic autoimmune diseases, such as systemic lupus erythematosus, etc.
  5. Patients with hypersensitivity to human or mouse monoclonal antibodies;
  6. Those who have a history of psychotropic drug abuse and cannot get rid of it or have mental disorders;
  7. According to the judgment of the researcher, there are serious concomitant diseases that endanger the patient's safety or affect the patient's ability to complete the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of translational treatment AE | up to 2 years
  Translational treatment-related AEs resulted in rates of surgery that were more than 30 days late or inoperable than originally planned
MPR | up to 2 years
  The proportion of patients whose primary tumor cell residual was less than 10% in the total number of patients enrolled after transformation therapy
pCR | up to 2 years
  Pathological complete response refers to that no tumor component or a small amount of carcinoma in situ component can be found on the horizontal line of pathological section after systemic treatment and surgical resection of the lesion.

SECONDARY OUTCOMES:
R0 resection rate | up to 2 years
  The proportion of patients who completed R0 resection through 3 cycles of immunotherapy combined with chemotherapy in the total enrolled population.R0 finger resection margin under microscope was negative.
Disease-free Survival，DFS | up to 2 years
  The time from randomization to disease recurrence or death due to disease progression

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Provincial People's Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xu T, Bai J, Zhao K, Chen X, Wang S, Zhu S, Sun C, Zhao C, Wang T, Zhu L, Hu M, Pang F, Zhang J, Wang W, Shu Y, Li F, Zhou Y. Induction Therapy of Tislelizumab Combined with Cisplatin and 5-Fluorouracil and Subsequent Conversion Surgery in Patients with Unresectable Advanced Esophageal Squamous Cell Carcinoma: A Phase 2, Single Center Study. Ann Surg Oncol. 2024 Dec;31(13):9321-9331. doi: 10.1245/s10434-024-16033-x. Epub 2024 Aug 23. PMID 39179863